CLINICAL TRIAL: NCT02985528
Title: Emergency Thoracic Ultrasound and Clinical Risk Management
Acronym: CLINRISKETUS
Status: Completed | Type: Observational
Sponsor: Guglielmo Trovato, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Guglielmo Trovato, MD, PhD, Professor of Medicine - Research Project Planning Unit, Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele
Organization: Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele (Other)
Other Study IDs: TUSMASTER
Record Dates: First submitted 2016-12-05; First posted 2016-12-07 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Chest Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- TUS positive: Ultrasound detection of pleuro-pulmonary disease and further diagnostic and imaging when needed
  Interventions: Other: further diagnostic
- CXR positive: Radiographic detection of pleuro-pulmonary disease and further diagnostic and imaging when needed
  Interventions: Other: further diagnostic

INTERVENTIONS:
Other: further diagnostic — further diagnostic procedures - mainly CHEST CT -
  Other Names: chest CT

SUMMARY:
Clinical risk assessment and management is mostly relevant in emergency. Thoracic ultrasound (TUS) has been proposed as an easy-option replacement for chest X-ray (CXR) in Emergency diagnosis of pneumonia, pleural effusion and pneumothorax. Investigators investigated CXR "unforeseen diagnosis", provided by TUS, exploring usefulness and sustainability of telementoring aimed at the management of clinical risk. This observational report includes a period of six months with a proactive concurrent adjunctive telementoring in TUS diagnosis using freely available smartphone applications for the transfer of images and movies.

DETAILED DESCRIPTION:
The present study describes a six months period of specialist activity of an Emergency Department physician. The aim is to display the performance in the subsets of difficult or unexpected thoracic ultrasound imaging performed by TUS, in a context with the prompt availability of all radiological facilities. The interaction of TUS telementoring, using WhatsApp® or Skype®, provided by another colleague, in another city and hospital, with a greater specific expertise in TUS, was devised to assure a concurrent mentorship by the School. This training has included a subsequent revaluation of clinical cases by the Ultrasound Course Lecturer in TUS and by the Director of the School of Clinical Ultrasound, with a reappraisal overview of all the available information. The approach was clinical and instrumental, and included:

A. clinical history; B. clinical examination of chest, neck, joints and abdomen; C. sequential ultrasound examination of the abdomen, thorax, pericardium; D. focus on pain symptoms: of chest, abdomen (with or without distention), lumbar region, neck; E. focus on dyspnea and/or cough and/or fever with detection of humid or dry lung sounds, chest dullness, of heart and/or pleura-pericardial sounds, and/or jugular congestion, checking also the mobility of the diaphragm and evaluating the collapsibility of the cava vein.

TUS was generally conducted with the patient in a sitting position, although the few patients (predominantly children), likely to experience severe discomfort during the procedure, were scanned in a semi-supine position. A systematic examination of all intercostal spaces was performed and TUS images, if present, were assessed for the number, location, shape, size, and breath-dependent changes in consolidation areas. Two main types of pattern of lung consolidation attributable to pneumonia were defined: hypoechoic consolidation and mixed consolidation. The presence of air bronchogram, fluid bronchogram, and basal pleural effusion was also reported. The size of the consolidation area was measured longitudinally and transversally, using the longest measurement, i.e., the maximal length of the consolidation area visible by TUS, for data analysis. For the purpose of this report, details on the measurements are not detailed.

The second opinion was provided outside the Hospital facility by a mentor (FMT), expert in Clinical Ultrasound, answering to the questions related to the images of videoclips of the actual patient in emergency. Images and movies were sent by WhatsApp. Reappraisal was performed subsequently, using all the available imaging - photos and videoclips, the clinical records and the outcome information, as obtainable by a short-term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in this study have satisfied one of these two criteria of unexpected diagnosis after TUS examination:

  1. Patients in which chest radiography was not diagnostic, or totally negative, in which thoracic ultrasound suggested evidence of a specific pathology (consolidation, effusion, pneumothorax), later confirmed by CT.
  2. Patients with detection of a chest disease on chest radiographs, and which a specific condition was further detailed, or differently addressed by the ultrasound procedure, and confirmed by CT.

Exclusion Criteria:

* patients with non-invasive pulse oximetry lower than 92.0% of Peripheral oxygen saturation (SpO2) , with clinical or instrumental signs of heart failure, in hemodialysis or with severe renal insufficiency, with a known diagnosis of solid or blood tumors.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: observations of a single physician of consecutivo emergency patients, (excluding trauma patients) addressed to a single facility for pain symptoms: of chest, abdomen (with or without distention), lumbar region, neck; and/or dyspnea and/or cough and/or fever with detection of humid or dry lung sounds, chest dullness, of heart and/or pleura-pericardial sounds, and/or jugular congestion.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
level of individual diagnostic accuracy of TUS vs. CXR | one day

IPD SHARING:
Plan to Share IPD: No